CLINICAL TRIAL: NCT05691374
Title: Evaluation of Functional and Biomechanical Outcome by Shear-wave Elastography in the Short to Intermediate Follow-up After Arthroscopic Rotator Cuff Repair
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-02061; mu23Mueller
Record Dates: First submitted 2023-01-10; First posted 2023-01-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Arthroscopic Rotator Cuff Repair (ARCR)
Keywords: shear-wave elastography (SWE); rotator cuff muscle; biceps muscle; deltoid muscle; trapezius muscle; functional outcome; biomechanical outcome; biceps tendon; infraspinatus muscle (ISP); teres minor muscle (TM); subscapularis muscle (SSC); supraspinatus muscle (SSP)
MeSH Terms: interventions — High-Energy Shock Waves; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ultrasound (US) examination — Shear-Wave Elastography (SWE) measurements of operated shoulder (quality, elasticity of repaired tendon) compared to healthy contralateral side. Parameters documented by regular US: Diameter of repaired tendon/ tendon thickness (mm), Rotator cuff muscle fatty infiltration (Grade 0-4), Signs of suture cut-through (yes | no), Signs of anchor displacement and location (lateral|medial row), Location of defect (at the foot print|medial cuff failure), Status of long biceps tendon (intact|in continuity|defect). Tissue elasticity measured by SWE in longitudinal orientation (in passive state and with active tension): Trapezius and Deltoid muscle: uninjured superficial muscle for individual patient muscle quality, SSP muscle and tendon: anterior and posterior part, SSC muscle and tendon: cranial and caudal part, ISP muscle and tendon, Biceps muscle and tendon: native (intraarticular) or subpectoral tenodesis (extraarticular)
Procedure: Clinical examination — Clinical examination for shoulder range of motion and strength measurement

SUMMARY:
This exploratory project will evaluate the biomechanical and functional intermediate-term outcome (2 to 5 years) after arthroscopic rotator cuff repair (ARCR) with modern non-invasive ultrasound techniques (especially shear wave elastography (SWE)), standardized physical examinations and patient-reported outcomes. It is to evaluate the biomechanical properties of tendons and muscles of the rotator cuff, as well as the biceps muscle after ARCR and to compare elasticity and structural properties to the healthy contralateral side.

DETAILED DESCRIPTION:
Arthroscopic repair of rotator cuff tears is commonly performed. However, recurrent tears after arthroscopic rotator cuff repair (ARCR) remain a significant clinical problem, especially in cases with large tears. Depending on literature, reported retear rates can range between 13% to 69%. Most likely, these tears reflect mechanical failure of the repair construct.

Ultrasound elastography is a recent technology and especially shear wave elastography (SWE) has experienced major developments in the past years. SWE offers an ultrasound based non-invasive quantitative tissue elasticity measurement by evaluating shear wave propagation speed which reflects the biomechanical properties of soft tissue. With this technique, the deltoid and trapezius muscle, several sections of the rotator cuff muscles and tendons as well as the proximal part of the long head of the biceps muscle can be evaluated. Results of the patient-reported outcomes and the physical examinations of the intermediate follow-up (2-5 years) will be compared with the data of the preoperative function.

It is a retrospective observational cohort study with additional prospective clinical data collection in terms of a physical examination and ultrasound examination.

There is no additional invasive procedure for this study.

ELIGIBILITY:
Inclusion Criteria:

* year of surgery between 2015 and 2020
* ARCR surgery in cases of:

  * Partial or complete supraspinatus (SSP) tear
  * Partial or complete supraspinatus (ISP) tear
  * Partial or complete subscapularis (SSC) tear
  * Combined SSP, ISP and SSC tear
* with or without biceps tenodesis during same procedure
* able to understand the content of the patient information / consent form and give consent to take part in the study

Exclusion Criteria:

* revision surgery (prior repair of the rotator cuff in the same shoulder)
* postoperative infections
* patients with a language barrier hindering questionnaire completion (either in German, French, Italian or English)
* legal incompetence
* not eligible for Ultrasound (BMI >35, persistent frozen shoulder)
* Prior surgery or injury of the contralateral shoulder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient selection from University Hospital Basel database
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Shear wave propagation velocity in kPa | one time assessment (at least 2 years postoperatively)
  Elasticity of tendon and muscle (shear wave propagation velocity in kPa)
Tendon integrity | one time assessment (at least 2 years postoperatively)
  Ultrasound of the repaired rotator cuff and biceps tendon (SSP, ISP, SSC, TM, long head of biceps)
Fatty infiltration (SSP, ISP, SSC, TM) | one time assessment (at least 2 years postoperatively)
  Fatty infiltration of the repaired rotator cuff (SSP, ISP, SSC, TM) by ultrasound
Diameter/Thickness of rotator cuff tendons (ISP, SSP, SSC, TM) | one time assessment (at least 2 years postoperatively)
  Diameter/Thickness of rotator cuff tendons (ISP, SSP, SSC, TM) by ultrasound
Status of implants e.g. anchors | one time assessment (at least 2 years postoperatively)
  Status of implants e.g. anchors by ultrasound
Suture cut-through (yes/no) | one time assessment (at least 2 years postoperatively)
  Suture cut-through (yes/no) by ultrasound

SECONDARY OUTCOMES:
Change in Constant Murley Score (CMS) | pre- operative, short-term (6 months postoperatively), and intermediate-term (at least 2 years) follow-up
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient after the treatment of a shoulder injury. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function.
Change in shoulder strength (kg) in 90° of abduction measured by handheld dynamometer | pre- operative, short-term (6 months postoperatively), and intermediate-term (at least 2 years) follow-up
  Change in shoulder strength (kg) in 90° of abduction measured by handheld dynamometer
Change in Patient-reported shoulder pain (NRS) | pre- operative, short-term (6 months postoperatively), and intermediate-term (at least 2 years) follow-up
  In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
Change in Patient-reported shoulder function (ASES) | pre- operative, short-term (6 months postoperatively), and intermediate-term (at least 2 years) follow-up
  The ASES is a 100-point scale that consists of two dimensions: pain and activities of daily living. There is one pain scale worth 50 points and ten activities of daily living worth 50 points. The pain score is calculated by subtracting the visual analogue scale (VAS) from 10 and multiplying it by 5. The 10 functional questions are scored on a 4-point scale (0-3) with a maximum functional score of 30.
Change in Subjective Shoulder Value (SSV) | pre- operative, short-term (6 months postoperatively), and intermediate-term (at least 2 years) follow-up
  The SSV score is defined as the subjective evaluation by the patient of shoulder function, expressed as a percentage of a normal shoulder. This score ranges from 0 to 100%.
Change in Quality of life assessed by EQ-5D-5- questionnaire | pre- operative, short-term (6 months postoperatively), and intermediate-term (at least 2 years) follow-up
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.The scale is numbered from 0 to 100. 100 means the best health you can imagine. 0 means the worst health you can imagine.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Müller, Prof. Dr. med., Study Director — University Hospital Basel, Department of Orthopaedic and Trauma surgery
Locations (1):
- University Hospital Basel, Department of Orthopaedic and Trauma surgery, Basel, Switzerland